CLINICAL TRIAL: NCT00329225
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Control, Clinical Evaluation of Insulin Plus Rosiglitazone (2mg and 4mg) Compared to Insulin Plus Placebo for 24 Weeks in Subjects With Type 2 Diabetes Mellitus Who Are Inadequately Controlled on Insulin
Brief Title: Rosiglitazone In Subjects With Type 2 Diabetes Mellitus Who Are Inadequately Controlled On Insulin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 49653/347; NCT00054782 (obsolete NCT alias)
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes Mellitus Thiazolidinediones Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: rosiglitazone

SUMMARY:
This 24-week study will compare the effects of adding the drug rosiglitazone (2mg and 4mg) or placebo to insulin in patients with Type 2 diabetes mellitus (non-insulin-dependent) who have not achieved their blood glucose goal using insulin alone. This study requires a total of seven visits during 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have Type II diabetes mellitus (non-insulin-dependent).
* Females must be post-menopausal (> 12 months without a menstrual period), surgically sterile, or must be using oral contraceptive, Norplant, Depo-provera, an IUD, or a diaphragm with spermicide or condoms. Females of childbearing potential must use acceptable contraceptive measures for at least one month prior to screening and for 30 days after completing the study.
* Must have been on insulin therapy alone continuously for at least 8 weeks prior to screening (minimum dose of 30 units per day). Patients taking insulin in combination with a single oral antidiabetic agent may have their oral agent discontinued and their insulin dose optimized over an 8 week period prior to screening if they are considered good study candidates in all other respects.
* HbA1c > 7.5% at Pre-screen or at Screen for subjects who discontinue their antidiabetic agent at pre-screening.
* Provide signed Informed Consent.

Exclusion Criteria:

* Females who are lactating, pregnant, or planning to become pregnant.
* Use of any drug called a thiazolidinedione within 6 months prior to screening, or more than one oral antidiabetic agent (including combinations of agents such as Glucovance) in combination with insulin in the 3 months prior to screening.
* Use of any investigational drug for blood glucose control within 3 months of screening regardless of the treatment regimen, or use of any other investigational agent within 30 days preceding study entry.
* Use of niacin (not including doses found in multivitamins) or oral corticosteroids within 3 months of screening.
* Patients with ongoing swelling due to fluid accumulation or history of such requiring treatment with a drug in the 12 months prior to screening.
* Patients with a documented history of significant hypersensitivity (e.g., difficulty swallowing, difficulty breathing, tachycardia or skin reaction) to the drugs called thiazolidinediones or similar drugs, or with prior fluid related intolerability to thiazolidinediones.
* Presence of clinically significant kidney or liver disease.
* Anemia.
* Presence of unstable or severe angina or coronary insufficiency.
* Patients with ongoing CHF (chronic heart failure) or history of CHF.
* Recent history or suspicion of current drug abuse or alcohol abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2002-09; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
HbA1c at each visit | 28 Weeks

SECONDARY OUTCOMES:
FPG at each visit C-peptide at each visit lipids at each visit BNP at each visit CRP at each visit PAI-1 at each visit MMP-9 at each visit | 28 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (111):
- United States (110):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Fairfield, Alabama
  - GSK Investigational Site, Fultondale, Alabama
  - GSK Investigational Site, Montgomery, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Concord, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Longmont, Colorado
  - GSK Investigational Site, Hamden, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Fort Meyers, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Gurnee, Illinois
  - GSK Investigational Site, Melrose Park, Illinois
  - GSK Investigational Site, Orland Park, Illinois
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Vernon Hills, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Madison, Kentucky
  - GSK Investigational Site, Lake Charles, Louisiana
  - GSK Investigational Site, Marrero, Louisiana
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Silver Spring, Maryland
  - GSK Investigational Site, Haverhill, Massachusetts
  - GSK Investigational Site, Taunton, Massachusetts
  - GSK Investigational Site, Cadillac, Michigan
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, Picayune, Mississippi
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Pahrump, Nevada
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Kenilworth, New Jersey
  - GSK Investigational Site, Martinsville, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Cooperstown, New York
  - GSK Investigational Site, Fulton, New York
  - GSK Investigational Site, Johnson City, New York
  - GSK Investigational Site, New Hyde Park, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Staten Island, New York
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Bismarck, North Dakota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Franklin, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Maumee, Ohio
  - GSK Investigational Site, Sidney, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Feasterville, Pennsylvania
  - GSK Investigational Site, Lansdale, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Reading, Pennsylvania
  - GSK Investigational Site, Scranton, Pennsylvania
  - GSK Investigational Site, Cranston, Rhode Island
  - GSK Investigational Site, Warick, Rhode Island
  - GSK Investigational Site, Summerville, South Carolina
  - GSK Investigational Site, Bartlett, Tennessee
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Cardova, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Chesapeake, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Federal Way, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- GSK Investigational Site

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Hollander P, Weston WM, Huang C, Chou H, and Porter LE. Low dose rosiglitazone significantly improves glycemic control without increasing adverse events in patients with T2DM not well controlled on insulin. Diabetes 2005;54(suppl 1):A3-4. Abstract 12-OR.
- [Derived] Hollander P, Yu D, Chou HS. Low-dose rosiglitazone in patients with insulin-requiring type 2 diabetes. Arch Intern Med. 2007 Jun 25;167(12):1284-90. doi: 10.1001/archinte.167.12.1284. PMID 17592102
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 49653/347 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 49653/347 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 49653/347 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 49653/347 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 49653/347 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 49653/347 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register